CLINICAL TRIAL: NCT02390466
Title: Multicentre, Open-label, Phase I/IIa Clinical Study of an Immunoprotective Therapeutic Vaccine Candidate (VAC-3S) in Human Immunodeficiency Virus Type 1 (HIV-1) Chronically Infected Patients Virologically Controlled on Antiretroviral Therapy (ART) Who Rose an Immune Response to VAC-3S During IVVAC-3S/P1
Brief Title: Open-label, Phase I/IIa Study of VAC-3S in HIV-1 Patients Who Showed an Immune Response to VAC-3S During IVVAC-3S/P1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InnaVirVax (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVVAC-3S/P2
Record Dates: First submitted 2015-01-30; First posted 2015-03-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2015-10

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VAC-3S (Experimental): 32µg/ml corresponding to 16µg/vaccination
  Interventions: Biological: VAC-3S

INTERVENTIONS:
Biological: VAC-3S — Administered via intra-muscular injection in the arm

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of VAC-3S in controlled HIV patients receiving standard of care antiretroviral treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patient,
* Age between 18 and 60 years,
* ART (Anti Retroviral Therapy) initiation ≥ 1 year ago,
* Plasma HIV RNA ≤ 200 copies/ml in the past 12 months,
* Plasma HIV RNA ≤ 50 copies/ml at the screening visit,
* CD4+ T cell count ≥ 200 cells/mm3,
* Nadir CD4+ T cell count ≥ 100 cells/mm3,
* Contraception in women with child-bearing potential,
* A total anti-3S titer ≥ 20 A.U. at any time point of IVVAC-3S/P1 clinical trial,
* Per protocol subject having completed the IVVAC-3S/P1 study.
* Patient affiliated to a social security system,
* Patient who has understood the protocol design and provided a signed written informed consent form,
* Patient who is willing and capable of cooperating to the extent and degree required by the protocol,
* Patient whom the investigator believes he/she can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits) and he/she will be available for all scheduled visits at the investigational site.

Exclusion Criteria:

* Administration of VAC-3S in the past year,
* Chronic active liver disease,
* History of HCV co-infection or ongoing replicating HCV (positive RT-PCR) or HBV (positive HbS Ag) coinfection,
* Any immunotherapy (e.g. IL-2, IL-7, growth hormone…) in the past year at the exception of VAC-3S,
* Any immunosuppressive therapy (glucocorticoids, cyclosporine, methotrexate) or chronic non-steroidal anti-inflammatory treatment in the past month,
* Ongoing pregnancy,
* Breastfeeding women,
* Patient with known sensitivities to investigational drug (see please the CIB),
* History of allergy to any vaccine,
* Any severe chronic condition that would interfere with the study,
* History of auto-immune disease,
* Organ transplant,
* Splenectomy,
* Psychiatric disorder significant enough to hinder participation as assessed by the investigator,
* Patient who has participated in a clinical research trial in the 30 days preceding the screening visit (V-1M-1).
* Patients with contraindications to intramuscular injections including, but not limited to, patients with thrombocytopenia and/or anomalies of the coagulation system,
* Any uncontrolled chronic or acute condition that in the opinion of the investigator would compromise the safety of the patient or the ability to properly administer the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients who tolerated 3 vaccinations with VAC-3S 16µg/mL at 4-weeks interval determined by safety parameter changes according to the DAIDS (Division of Acquired Immunodeficiency Syndrome) Adverse Events (AE) Grading Table. | From Day 0 to week 16

SECONDARY OUTCOMES:
Number of patients who tolerated a fourth booster injection of VAC-3S 16µg/mL determined by safety parameter changes according to the DAIDS (Division of Acquired Immunodeficiency Syndrome) Adverse Events (AE) Grading Table. | From Week 16 to Week 48
Anti-3S antibody titers | From Day 0 to Week 48
Markers of progression to AIDS. Markers include CD4+ cell count, viral load, and phenotypic markers of lymphocyte differentiation and activation | From Day 0 to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Ho Tsong Fang, DVM PhD, Study Director — InnaVirVax
Locations (2):
- France (2):
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Cochin Saint Vincent de Paul, Paris